CLINICAL TRIAL: NCT06876792
Title: Electrical Impedance Tomography-Derived Flow Index for Predicting Weaning Success and Post-Extubation Outcomes: A Multicenter Prospective Observational Study
Acronym: EIT-FI Weaning
Status: Completed | Type: Observational
Sponsor: Ruijin Hospital (Other)
Collaborators: Shanghai Rui Jin Hospital (Unknown); Foshan Hospital of Traditional Chinese Medicine (Other); Fujian Provincial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202530
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Respiratory Drive; Acute Respiratory Failure
Keywords: acute respiratory failure; Respiratory drive; Electrical Impedance Tomography (EIT); ventilator weaning; spontaneous breathing trial; pendelluft; patient self-inflicted lung injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Conventional method Respiratory Drive group: Conventional method Respiratory Drive group（Methods include: esophageal pressure monitoring, airway obstruction pressure (P0.1) )
  Interventions: Device: electrical impedance tomography

INTERVENTIONS:
Device: electrical impedance tomography — Respiratory drive assessed by flow index measured by electrical impedance tomography.

SUMMARY:
Accurate prediction of readiness to liberate patients from mechanical ventilation remains challenging. Conventional indices such as the rapid shallow breathing index (RSBI) and maximal inspiratory pressure (MIP) often miss early signs of injurious breathing patterns or regional ventilation asynchrony that can lead to extubation failure. Electrical impedance tomography (EIT) provides continuous, non-invasive imaging of regional lung ventilation. We developed a novel EIT-derived Flow Index (FI) which integrates the magnitude of inspiratory effort with the temporal synchrony of lung filling. This prospective, multicenter observational study aimed to (1) validate the predictive value of FI during spontaneous breathing trials (SBT) compared with conventional weaning indices, and (2) investigate the association between FI and pendelluft magnitude as a potential marker of patient self-inflicted lung injury (P-SILI).

DETAILED DESCRIPTION:
This multicenter observational study was conducted in three ICUs in China. Adult patients (≥18 years) who received invasive mechanical ventilation for

≥48 hours and met standard criteria for SBT readiness underwent a standardized 30-minute pressure-support SBT (PSV 8 cmH₂O, PEEP 5 cmH₂O, FiO₂ ≤0.5). Continuous EIT recordings were performed to calculate global and regional FI from pixel-level inspiratory flow-time curves. Pendelluft magnitude was quantified as the percentage of intrapulmonary gas redistribution during inspiration. Conventional indices (RSBI, MIP, P0.1, NIF) and physiological variables were recorded. Primary Endpoint: SBT success (completion without respiratory distress, desaturation, or hemodynamic instability).

Secondary Endpoints:

* Reintubation within 48 h
* Weaning failure
* Ventilator-free days at day 7
* ICU mortality Predictive accuracy was evaluated via ROC analysis in training (n=90) and validation (n=60) cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Acute respiratory failure requiring intubation and mechanical ventilation ≥48 hours
* Hemodynamic stability (no escalation of vasoactive agents)
* Oxygenation: FiO₂ ≤0.5, PEEP ≤8 cmH₂O
* Meeting standard ICU criteria for SBT readiness

Exclusion Criteria:

* Neuromuscular diseases impairing spontaneous breathing
* High cervical spinal cord injury
* Deep sedation (RASS ≤-3)
* Inadequate EIT signal quality
* Contraindications to EIT (e.g., implanted cardiac devices)
* Pregnancy
* Expected survival <24 h

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. 150 critically ill patients requiring respiratory support were planned for inclusion
  2. Age ≥18 years
  3. Gender is not limited
  4. Patients with expected duration of respiratory support >24 hours
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Spontaneous Breathing Trial (SBT) Success Rate | Within 30 minutes of Spontaneous Breathing Trial (SBT)
  Proportion of patients who complete the 30-minute Spontaneous Breathing Trial (SBT) without signs of respiratory distress, desaturation, or hemodynamic instability.

SECONDARY OUTCOMES:
Reintubation Rate within 48 hours | Within 48 hours after extubation.
  Proportion of patients requiring reintubation within 48 hours following successful extubation.
Ventilator-Free Days by Day 7 | Within 7 days after extubation.
  Number of days free from mechanical ventilation within 7 days after extubation.
ICU Mortality | during the ICU stay or within 24 hours following transfer out of the ICU
  Mortality rate of patients during their ICU stay in this study.
Correlation between FI and pendelluff magnitude | During the 30-minute SBT.
  Pearson correlation coefficient between the Flow Index (FI) and pendelluff magnitude.
Predictive value of FI vs. RSBI, MIP, P0.1 for SBT success | During the 30-minute SBT.
  Comparison of the area under the ROC curve (AUC) for FI and conventional indices (RSBI, MIP, P0.1) in predicting SBT success.

CONTACTS AND LOCATIONS:
Overall Officials: Hongping Qu, Study Chair — Department of Critical Care Medicine，Ruijin Hospital，Shanghai Jiao Tong University School of Medicine; Jialin Liu, Study Director — Department of Critical Care Medicine，Ruijin Hospital，Shanghai Jiao Tong University School of Medicine; rui zhang, Principal Investigator — Department of Critical Care Medicine，Ruijin Hospital，Shanghai Jiao Tong University School of Medicine
Locations (3):
- China (3):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - Department of Critical Care Medicine，Ruijin Hospital，Shanghai Jiao Tong University School of Medicine，Shanghai，China., Shanghai

IPD SHARING:
Plan to Share IPD: No